CLINICAL TRIAL: NCT07149974
Title: Developing an EEG-fNIRS Neurofeedback Application for Brain Training for Autistic Children
Brief Title: Neurofeedback Training for Autistic Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: HOME Psychological Services Ltd. (Unknown); ANT Asia Pacific (Unknown)
Responsible Party: Principal Investigator, YEUNG Kin Chung Michael, Assistant professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-2023-0505; ITS/077/22 (Other Grant/Funding Number: Innovation and Technology Commission)
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Autism; Autistic Disorders Spectrum; Neurofeedback; EEG; fNIRS
Keywords: ASD; Autistic; Neurofeedback; EEG; fNIRS
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: The participants will be randomly and equally assigned to one of three neurofeedback training groups: (1) Combined EEG-fNIRS, (2) EEG, and (3) fNIRS. Each participant will complete a neurophysiological assessment (1) before and (2) immediately after a 12-session program (two 1-hour sessions per week).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During each training session, a cap adjusted to the participant's head size will be used to mount the EEG and fNIRS sensors. The hardware setup will be the same for all groups to ensure that both the participant and experimenter are blinded to the training group. Besides, all participants will be identified by numbers, which are randomly assigned to one of three conditions by the Principal Investigator, who does not involve in either the assessment or training session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined EEG-fNIRS group (Experimental): The participants will undertake two essential phases of neurofeedback training: (1) baseline and (2) training. During baseline phase (typically 3 minutes), the user plays the default neurofeedback game to obtain baseline EEG and fNIRS recordings. On the basis of these signals, the mean and standard deviation of the index of interest will be extracted and calculated. During the training phase (typically 5 minutes), the signal processing is almost identical to the one during baseline phase, but the moment-to-moment outcome variable will be Z-normalized according to the mean and SD of the target index. Once the data is pushed to the LSL stream for use in neurofeedback game interaction, participants can see the corresponding changes in the game screen. For the combined EEG-fNIRS group, both the EEG and fNIRS indices will be be extracted. To encourage integration, the lower value of the two will be chosen as the outcome variable.
  Interventions: Device: EEG and fNIRS
- EEG group (Experimental): The participants will undertake two essential phases of neurofeedback training: (1) baseline and (2) training. During baseline phase (typically 3 minutes), the user plays the default neurofeedback game to obtain baseline EEG and fNIRS recordings. On the basis of these signals, the mean and standard deviation of the index of interest will be extracted and calculated. During the training phase (typically 5 minutes), the signal processing is almost identical to the one during baseline phase, but the moment-to-moment outcome variable will be Z-normalized according to the mean and SD of the target index. Once the data is pushed to the LSL stream for use in neurofeedback game interaction, participants can see the corresponding changes in the game screen. For EEG, the frontal theta/beta ratio, left-right difference in frontal alpha power, and the mu power are chosen as the target training indices.
  Interventions: Device: EEG
- fNIRS group (Experimental): The participants will undertake two essential phases of neurofeedback training: (1) baseline and (2) training. During baseline phase (typically 3 minutes), the user plays the default neurofeedback game to obtain baseline EEG and fNIRS recordings. On the basis of these signals, the mean and standard deviation of the index of interest will be extracted and calculated. During the training phase (typically 5 minutes), the signal processing is almost identical to the one during baseline phase, but the moment-to-moment outcome variable will be Z-normalized according to the mean and SD of the target index. Once the data is pushed to the LSL stream for use in neurofeedback game interaction, participants can see the corresponding changes in the game screen. For fNIRS, the level of prefrontal activation (HbO or HbR), the left-right difference in prefrontal activation, and the motor cortex activation are chosen as the target training indices, respectively.
  Interventions: Device: fNIRS

INTERVENTIONS:
Device: EEG and fNIRS — For EEG and fNIRS, EEG signals will be recorded using the ANT Neuro eego rt 8 amplifier device (ANT Neuro, Hengelo, The Netherlands), with electrodes placed at C3, C4, F3, F4, Fpz, M1, M2, and GND (ground). fNIRS signals will be recorded using the Artinis Brite Lite fNIRS device(Artinis Medical Systems, The Netherlands). The overall channel configuration consists of eight sources and four detectors. Among these, four sources (T2a-d) and four detectors (R1-4) form four short-separation channels, while the remaining four sources and four detectors constitute six long-separation channels (T1-R1, T3-R1, T3-R2, T4-R3, T5-R3, T5-R4). The overall configuration is approximately arranged in two L-shaped layouts surrounding the F3 and F4 regions.
  Arms: Combined EEG-fNIRS group
Device: EEG — EEG signals will be recorded using the ANT Neuro eego rt 8 amplifier device (ANT Neuro, Hengelo, The Netherlands), with electrodes placed at C3, C4, F3, F4, Fpz, M1, M2, and GND (ground).
  Arms: EEG group
Device: fNIRS — fNIRS signals will be recorded using the Artinis Brite Lite fNIRS device(Artinis Medical Systems, The Netherlands). The overall channel configuration consists of eight sources and four detectors. Among these, four sources (T2a-d) and four detectors (R1-4) form four short-separation channels, while the remaining four sources and four detectors constitute six long-separation channels (T1-R1, T3-R1, T3-R2, T4-R3, T5-R3, T5-R4). The overall configuration is approximately arranged in two L-shaped layouts surrounding the F3 and F4 regions.
  Arms: fNIRS group

SUMMARY:
The goal of this study is to learn if a new brain training method, called combined electroencephalography (EEG) and functional near-infrared spectroscopy (fNIRS) neurofeedback, can improve thinking, emotions, and social functioning in children with autism spectrum disorder (ASD). It will also learn if this training is practical and safe to use with children in Hong Kong.

The main questions this study aims to answer are:

* Does combined EEG-fNIRS neurofeedback improve attention, emotion regulation, and social skills in children with ASD?
* Is this type of neurofeedback training feasible and well-tolerated by children? Researchers will compare the new combined EEG-fNIRS training with single EEG or fNIRS training to see if it provides additional benefits.

Participants will:

.Receive sessions of EEG-fNIRS neurofeedback training. .Complete assessments of thinking skills, emotional regulation, and social functioning before and after training.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a lifelong neurodevelopmental condition characterized by difficulties in social communication and interaction, often accompanied by cognitive and emotional regulation challenges. In Hong Kong and many other countries, ASD is increasingly prevalent. Despite this, the brain health of autistic individuals has been relatively neglected in both healthcare systems and public policies. There is also a lack of approaches and technologies that directly intervene with brain function. Since many autistic children experience poor vocational and health outcomes in adulthood, there is a strong need to develop effective and accessible neuroscience-based treatments.

This project aims to apply cutting-edge neuroscientific methods to develop an innovative closed-loop brain training intervention for children with ASD. The intervention will combine electroencephalography (EEG) and functional near-infrared spectroscopy (fNIRS) in a unified neurofeedback training system. Neurofeedback training teaches individuals to self-regulate brain activity by providing real-time feedback. In the traditional neurofeedback study, EEG has been used to guide neurofeedback by monitoring electrical activity in the brain, while more recently fNIRS has been used to track hemodynamic activity. However, no existing neurofeedback system has integrated these two modalities. Combining EEG and fNIRS provides an opportunity to enhance neurovascular coupling, the relationship between neural activity and blood flow, which is often altered in neuropsychiatric conditions such as autism.

The proposed neurofeedback application will include multiple training modules designed to address cognitive, emotional, and social difficulties common in autism. The cognitive training module will target brain activity patterns associated with attention and executive function. The affective training module will focus on modulating frontal brain activity linked to emotional regulation. The social training module will aim to enhance neural and hemodynamic activity associated with social cognition and communication. By integrating both EEG and fNIRS indices, the system will encourage children to regulate electrical and hemodynamic activity simultaneously, which cannot be achieved using either modality alone.

To maximize engagement, the application will incorporate ecologically valid feedback stimuli and reward-based learning principles. Instead of relying solely on abstract indicators such as bars or tones, the feedback will involve intrinsically rewarding stimuli, such as videos or positive visual cues, to increase motivation and adherence. The training difficulty will be adjusted progressively based on individual performance to ensure sustained engagement and improvement.

In addition, the system will be developed as a cross-device application using open-source lab streaming layer (LSL) software, ensuring compatibility with a wide range of EEG and fNIRS devices. The hardware and software will be optimized to ensure high-quality signals, including the use of shielded wet electrodes for EEG to reduce noise and short-separation channels in fNIRS to minimize extracerebral signal contamination. These features will allow neurofeedback training to be conducted with minimal environmental interference, enhancing both reliability and clinical applicability.

Through this proof-of-concept project, this project aims to establish the feasibility of combined EEG-fNIRS neurofeedback as a novel form of brain training for autistic children. If successful, this approach has the potential to offer a comprehensive, technology-based neurorehabilitation solution that can improve functional outcomes, reduce healthcare burdens, and foster innovation in neurotechnology in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 12 years
* Previous diagnosis of autism spectrum disorder (ASD) or Asperger's syndrome
* No intellectual impairment or studying in mainstream schools
* Right-handedness
* Normal or corrected-to-normal vision

Exclusion Criteria:

- Not meeting any of the above inclusion criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of treatments for autistic individuals | Within 1 week before the first training session, and within 1 week after the last training session
  The Autism Treatment Evaluation Checklist (ATEC) assesses the effectiveness of treatments for autistic individuals. It is completed by parent and consists of four subscales in different aspects of functioning, including Speech/Language/Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior. Parents are required to answer each question using a 3-point scale ranging from 0 (not true) to 2 (true). The checklist can typically be completed in about 5 minutes.
Social behavior and Social impairments | Within 1 week before the first training session, and within 1 week after the last training session
  The Social Responsiveness Scale, Second Edition (SRS-2) is a 65-item questionnaire designed to assess social behavior and identify social impairments associated with autism spectrum disorders. It is completed by parent and evaluates 5 subscales, including social awareness, social cognition, social communication, social motivation, and restricted interests and repetitive behaviors. Respondents rate each item on a 4-point Likert scale, ranging from 0 (not true) to 3 (always true), reflecting the frequency and severity of observed behaviors. The questionnaire can typically be completed in around 10 minutes.
Executive function in children and adolescents | Within 1 week before the first training session, and within 1 week after the last training session
  The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) is a 63-item questionnaire designed to assess executive function in children and adolescents. It is completed by parent and evaluates subscales such as behavioral regulation, emotional control, and cognitive processes. Respondents rate each item on a 3-point scale ranging from 1 (never) to 3 (often), indicating the frequency of behaviors. The questionnaire can typically be completed in around 15 minutes.
Anxiety and depression symptoms in children and adolescents | Within 1 week before the first training session, and within 1 week after the last training session
  The Revised Children's Anxiety and Depression Scale-Parent Version (RCADS-P) is a 25-item questionnaire designed to assess anxiety and depression symptoms in children and adolescents. Completed by parent, it evaluates key emotional domains, including generalized anxiety, panic disorder, separation anxiety, social phobia, obsessive-compulsive disorder, and major depressive disorder. Parents rate each item based on their child's recent behavior using a 4-point Likert scale: 0 (never), 1 (sometimes), 2 (often), and 3 (always), reflecting the frequency of symptoms. The checklist can typically be completed in around 3 minutes.

SECONDARY OUTCOMES:
Go/No-go(post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Go/No-go mean reaction time
Go/No-go (post; Accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Go/No-go accuracy
Sternberg Working Memory Task (post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Sternberg task mean reaction time
Sternberg Working Memory Task (post; Accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Sternberg task accuracy
Task Switching (post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Task Switching mean reaction time
Task Switching (post; Accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Task Switching accuracy
Child Eyes Test (post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Child Eyes Test mean reaction time
Child Eyes Test (post; Accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Child Eyes Test accuracy
Facial Emotion Recognition Task (post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Facial Emotion Recognition mean reaction time
Facial Emotion Recognition Task (post; Accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Facial Emotion Recognition accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Kin Chung Michael Yeung, PhD, Principal Investigator — Education University of Hong Kong
Locations (1):
- Faculty of Education And Human Development OF The Educational University Of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
All data related to this study will be kept strictly confidential and will be accessible only to the research team for research purposes. Study findings may be published in academic journals or presented at conferences; however, the names of participants and their families will remain confidential. All assessment instruments will be identified by coded numbers rather than names, and all personal information will be stored in a locked filing cabinet until the fifth year following the dissemination of study results. The Confidentiality and Privacy Ordinance of The Educational University Of Hong Kong shall protect and keep all medical data.

REFERENCES:
- [Background] Wang SY, Lin IM, Fan SY, Tsai YC, Yen CF, Yeh YC, Huang MF, Lee Y, Chiu NM, Hung CF, Wang PW, Liu TL, Lin HC. The effects of alpha asymmetry and high-beta down-training neurofeedback for patients with the major depressive disorder and anxiety symptoms. J Affect Disord. 2019 Oct 1;257:287-296. doi: 10.1016/j.jad.2019.07.026. Epub 2019 Jul 5. PMID 31302517
- [Background] Van Doren J, Arns M, Heinrich H, Vollebregt MA, Strehl U, K Loo S. Sustained effects of neurofeedback in ADHD: a systematic review and meta-analysis. Eur Child Adolesc Psychiatry. 2019 Mar;28(3):293-305. doi: 10.1007/s00787-018-1121-4. Epub 2018 Feb 14. PMID 29445867
- [Background] Trambaiolli LR, Kohl SH, Linden DEJ, Mehler DMA. Neurofeedback training in major depressive disorder: A systematic review of clinical efficacy, study quality and reporting practices. Neurosci Biobehav Rev. 2021 Jun;125:33-56. doi: 10.1016/j.neubiorev.2021.02.015. Epub 2021 Feb 12. PMID 33587957
- [Background] The Government of the Hong Kong Special Administrative Region. (2019). EDB to enhance support for students with autism spectrum disorders. Retrieved August 24, 2022, from https://www.info.gov.hk/gia/general/201910/03/P2019100300291.htm?fontSize=1.
- [Background] Steingrimsson S, Bilonic G, Ekelund AC, Larson T, Stadig I, Svensson M, Vukovic IS, Wartenberg C, Wrede O, Bernhardsson S. Electroencephalography-based neurofeedback as treatment for post-traumatic stress disorder: A systematic review and meta-analysis. Eur Psychiatry. 2020 Jan 31;63(1):e7. doi: 10.1192/j.eurpsy.2019.7. PMID 32093790
- [Background] Shaffer RC, Pedapati EV, Shic F, Gaietto K, Bowers K, Wink LK, Erickson CA. Brief Report: Diminished Gaze Preference for Dynamic Social Interaction Scenes in Youth with Autism Spectrum Disorders. J Autism Dev Disord. 2017 Feb;47(2):506-513. doi: 10.1007/s10803-016-2975-2. PMID 27878742
- [Background] Russo, G. M., Balkin, R. S., & Lenz, A. S. (2022). A meta-analysis of neurofeedback for treating anxiety-spectrum disorders. Journal of Counseling & Development, 100(3), 236-251.
- [Background] Rosson S, de Filippis R, Croatto G, Collantoni E, Pallottino S, Guinart D, Brunoni AR, Dell'Osso B, Pigato G, Hyde J, Brandt V, Cortese S, Fiedorowicz JG, Petrides G, Correll CU, Solmi M. Brain stimulation and other biological non-pharmacological interventions in mental disorders: An umbrella review. Neurosci Biobehav Rev. 2022 Aug;139:104743. doi: 10.1016/j.neubiorev.2022.104743. Epub 2022 Jun 14. PMID 35714757
- [Background] Pineda JA, Carrasco K, Datko M, Pillen S, Schalles M. Neurofeedback training produces normalization in behavioural and electrophysiological measures of high-functioning autism. Philos Trans R Soc Lond B Biol Sci. 2014 Apr 28;369(1644):20130183. doi: 10.1098/rstb.2013.0183. Print 2014. PMID 24778378
- [Background] Pineda, J. A., Brang, D., Hecht, E., Edwards, L., Carey, S., Bacon, M., ... & Rork, A. (2008). Positive behavioral and electrophysiological changes following neurofeedback training in children with autism. Research in Autism Spectrum Disorders, 2(3), 557-581.
- [Background] Perihan C, Burke M, Bowman-Perrott L, Bicer A, Gallup J, Thompson J, Sallese M. Effects of Cognitive Behavioral Therapy for Reducing Anxiety in Children with High Functioning ASD: A Systematic Review and Meta-Analysis. J Autism Dev Disord. 2020 Jun;50(6):1958-1972. doi: 10.1007/s10803-019-03949-7. PMID 30810842
- [Background] Mehler DMA, Sokunbi MO, Habes I, Barawi K, Subramanian L, Range M, Evans J, Hood K, Luhrs M, Keedwell P, Goebel R, Linden DEJ. Targeting the affective brain-a randomized controlled trial of real-time fMRI neurofeedback in patients with depression. Neuropsychopharmacology. 2018 Dec;43(13):2578-2585. doi: 10.1038/s41386-018-0126-5. Epub 2018 Jun 23. PMID 29967368
- [Background] Marzbani H, Marateb HR, Mansourian M. Neurofeedback: A Comprehensive Review on System Design, Methodology and Clinical Applications. Basic Clin Neurosci. 2016 Apr;7(2):143-58. doi: 10.15412/J.BCN.03070208. PMID 27303609
- [Background] Marx AM, Ehlis AC, Furdea A, Holtmann M, Banaschewski T, Brandeis D, Rothenberger A, Gevensleben H, Freitag CM, Fuchsenberger Y, Fallgatter AJ, Strehl U. Near-infrared spectroscopy (NIRS) neurofeedback as a treatment for children with attention deficit hyperactivity disorder (ADHD)-a pilot study. Front Hum Neurosci. 2015 Jan 7;8:1038. doi: 10.3389/fnhum.2014.01038. eCollection 2014. PMID 25610390
- [Background] Llorente AM, Voigt RG, Williams J, Frailey JK, Satz P, D'Elia LF. Children's Color Trails Test 1 & 2: test-retest reliability and factorial validity. Clin Neuropsychol. 2009 May;23(4):645-60. doi: 10.1080/13854040802427795. Epub 2008 Oct 21. PMID 18942031
- [Background] Liu, Z., Shore, J., Wang, M., Yuan, F., Buss, A., & Zhao, X. (2021). A systematic review on hybrid EEG/fNIRS in brain-computer interface. Biomedical Signal Processing and Control, 68, 102595.
- [Background] Li K, Jiang Y, Gong Y, Zhao W, Zhao Z, Liu X, Kendrick KM, Zhu C, Becker B. Functional near-infrared spectroscopy-informed neurofeedback: regional-specific modulation of lateral orbitofrontal activation and cognitive flexibility. Neurophotonics. 2019 Apr;6(2):025011. doi: 10.1117/1.NPh.6.2.025011. Epub 2019 Jun 8. PMID 31930153
- [Background] Kouijzer, M. E., de Moor, J. M., Gerrits, B. J., Congedo, M., & van Schie, H. T. (2009). Neurofeedback improves executive functioning in children with autism spectrum disorders. Research in Autism Spectrum Disorders, 3(1), 145-162.
- [Background] Kothe C, Shirazi SY, Stenner T, Medine D, Boulay C, Grivich MI, Artoni F, Mullen T, Delorme A, Makeig S. The Lab Streaming Layer for Synchronized Multimodal Recording. bioRxiv [Preprint]. 2025 Jul 14:2024.02.13.580071. doi: 10.1101/2024.02.13.580071. PMID 38405712
- [Background] Kober SE, Spork R, Bauernfeind G, Wood G. Age-related differences in the within-session trainability of hemodynamic parameters: a near-infrared spectroscopy-based neurofeedback study. Neurobiol Aging. 2019 Sep;81:127-137. doi: 10.1016/j.neurobiolaging.2019.05.022. Epub 2019 Jun 5. PMID 31280116
- [Background] Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb;5(2):e45. doi: 10.1371/journal.pmed.0050045. PMID 18303940
- [Background] Kimmig AS, Dresler T, Hudak J, Haeussinger FB, Wildgruber D, Fallgatter AJ, Ehlis AC, Kreifelts B. Feasibility of NIRS-based neurofeedback training in social anxiety disorder: behavioral and neural correlates. J Neural Transm (Vienna). 2019 Sep;126(9):1175-1185. doi: 10.1007/s00702-018-1954-5. Epub 2018 Nov 29. PMID 30498952
- [Background] Kellems, R. O., Charlton, C. T., Black, B., Bussey, H., Ferguson, R., Gonçalves, B. F., ... & Vallejo, S. (2022). Social Engagement of Elementary-Aged Children With Autism Live Animation Avatar Versus Human Interaction. Journal of Special Education Technology, 01626434221094792.
- [Background] Hammond DC. Neurofeedback with anxiety and affective disorders. Child Adolesc Psychiatr Clin N Am. 2005 Jan;14(1):105-23, vii. doi: 10.1016/j.chc.2004.07.008. PMID 15564054
- [Background] Guven A, Altinkaynak M, Dolu N, Demirci E, Ozmen S, Izzetoglu M, Pektas F. Effects of Methylphenidate on Reaction Time in Children with Attention Deficit / Hyperactivity Disorder. Noro Psikiyatr Ars. 2019 Mar;56(1):27-31. doi: 10.29399/npa.22873. Epub 2018 Apr 20. PMID 30911234
- [Background] Friedrich EV, Sivanathan A, Lim T, Suttie N, Louchart S, Pillen S, Pineda JA. An Effective Neurofeedback Intervention to Improve Social Interactions in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2015 Dec;45(12):4084-100. doi: 10.1007/s10803-015-2523-5. PMID 26210513
- [Background] Fernandez-Alvarez J, Grassi M, Colombo D, Botella C, Cipresso P, Perna G, Riva G. Efficacy of bio- and neurofeedback for depression: a meta-analysis. Psychol Med. 2022 Jan;52(2):201-216. doi: 10.1017/S0033291721004396. Epub 2021 Nov 15. PMID 34776024
- [Background] Ehlis, A. C., Barth, B., Hudak, J., Storchak, H., Weber, L., Kimmig, A. C. S., ... & Fallgatter, A. J. (2018). Near-infrared spectroscopy as a new tool for neurofeedback training: Applications in psychiatry and methodological considerations. Japanese Psychological Research, 60(4), 225-241.
- [Background] Demetriou EA, Lampit A, Quintana DS, Naismith SL, Song YJC, Pye JE, Hickie I, Guastella AJ. Autism spectrum disorders: a meta-analysis of executive function. Mol Psychiatry. 2018 May;23(5):1198-1204. doi: 10.1038/mp.2017.75. Epub 2017 Apr 25. PMID 28439105
- [Background] Danial JT, Wood JJ. Cognitive behavioral therapy for children with autism: review and considerations for future research. J Dev Behav Pediatr. 2013 Nov-Dec;34(9):702-15. doi: 10.1097/DBP.0b013e31829f676c. PMID 23917373
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Arns M, de Ridder S, Strehl U, Breteler M, Coenen A. Efficacy of neurofeedback treatment in ADHD: the effects on inattention, impulsivity and hyperactivity: a meta-analysis. Clin EEG Neurosci. 2009 Jul;40(3):180-9. doi: 10.1177/155005940904000311. PMID 19715181
- [Background] American Psychiatric Association (2022). Diagnostic and statistical manual of mental disorders (5th Edition, Text Revision). Washington, D.C.: American Psychiatric Publishing.